CLINICAL TRIAL: NCT00808405
Title: Prospective Study of Pharmacokinetics, Clinical and Virologic Response to Acyclovir Episodic Therapy for Genital Herpes Ulcers in HIV Negative African Women
Brief Title: GUD Clinical and Virologic Response to Acyclovir in HIV Negative African Women
Acronym: PK/GUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Connie Celum, MPH/ Principal Investigator, Protocol Co-Chair, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34708-A; U01AI052054 (NIH)
Record Dates: First submitted 2008-11-25; First posted 2008-12-15 (Estimated); Results first posted 2012-05-18 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-11

CONDITIONS: Genital Herpes
Keywords: herpes simplex virus; acyclovir; HSV shedding; women; Africa
MeSH Terms: conditions — Herpes Genitalis; Herpes Simplex | interventions — Acyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- acyclovir (Active Comparator)
  Interventions: Drug: acyclovir
- placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: acyclovir — 400mg taken orally three times daily for 5 days
  Arms: acyclovir
Drug: matching placebo — matching placebo taken orally three times daily for 5 days.
  Arms: placebo

SUMMARY:
To examine the time to healing of genital lesion and duration of herpes simplex virus (HSV) shedding from genetic ulcer disease (GUD) among 90 HIV-negative African women who have a history of GUD and are HSV-2 seropositive and HIV-1 seronegative randomized in a 2:1 ratio to receive episodic acyclovir 400mg orally three times daily or matching placebo three times daily for 5 days and who are followed for a total of 13 days.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative as determined by concordant rapid testing
* HSV-2 seropositive (Focus HerpeSelect >3.4)
* At least one prior occurrence of GUD
* 18-50 years of age

Exclusion Criteria:

* Current use, or use w/in past 7 days of acyclovir, valacyclovir, or famciclovir
* Prior hypersensitivity &/or allergic reaction to acyclovir
* Use of probenicid
* Current use, or use within past 28 days, of an investigational agent
* Currently pregnant or nursing
* Currently plan to become pregnant during next 3 months
* Any condition that will interfere with successful completion of study procedures

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington; Anna Wald, MD, MPH, Principal Investigator — University of Washington
Locations (2):
- Reproductive Health and HIV Research Unit (RHRU), Johannesburg, South Africa
- Center for Infectious Disease Research of Zambia (CIDRZ), Lusaka, Zambia

REFERENCES:
- [Background] Celum C, Wald A, Hughes J, Sanchez J, Reid S, Delany-Moretlwe S, Cowan F, Casapia M, Ortiz A, Fuchs J, Buchbinder S, Koblin B, Zwerski S, Rose S, Wang J, Corey L; HPTN 039 Protocol Team. Effect of aciclovir on HIV-1 acquisition in herpes simplex virus 2 seropositive women and men who have sex with men: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Jun 21;371(9630):2109-19. doi: 10.1016/S0140-6736(08)60920-4. PMID 18572080
- [Background] Lu Y, Celum C, Wald A, Baeten JM, Cowan F, Delany-Moretlwe S, Reid SE, Hughes JP, Wilcox E, Corey L, Hendrix CW. Acyclovir achieves a lower concentration in African HIV-seronegative, herpes simplex virus 2-seropositive women than in non-African populations. Antimicrob Agents Chemother. 2012 May;56(5):2777-9. doi: 10.1128/AAC.06160-11. Epub 2012 Feb 13. PMID 22330926
- [Derived] Baeten JM, Reid SE, Delany-Moretlwe S, Hughes JP, Wang RS, Wilcox E, Limbada M, Akpomiemie G, Corey L, Wald A, Celum C. Clinical and virologic response to episodic acyclovir for genital ulcers among HIV-1 seronegative, herpes simplex virus type 2 seropositive African women: a randomized, placebo-controlled trial. Sex Transm Dis. 2012 Jan;39(1):21-4. doi: 10.1097/OLQ.0b013e31823b50c6. PMID 22183840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January and December 2009, women from Johannesburg, South Africa and Lusaka, Zambia who had previously participated in the HPTN 039 (NCT00076232) study, as well as other women in the community who presented to the research clinics with genetic ulcer disease (GUD) during the recruitment period, were invited to participate in the study.
Groups:
- Acyclovir: Acyclovir 400 mg orally three times daily
- Placebo: Matching placebo tablet
Period: Overall Study
Arm/Group | Acyclovir | Placebo
Started | 61 | 27
Completed | 61 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acyclovir | Placebo | Total
Number analyzed (Participants) | 61 | 27 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 27 | 88
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.66 (10.28) | 38.15 (10.31) | 38.5 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 27 | 88
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Zambia | 31 | 13 | 44
  South Africa | 30 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Time to Healing of Genital Lesions
Description: To examine time to healing of genital lesions among women who have a history of GUD and are HSV-2 seropositive and HIV-1 seronegative, and who are randomized to 400mg acyclovir or matching placebo
Time Frame: Days 1-5, 7, 9, 11, 13
Population: Eligible women were 18-50 years of age, HIV-1 seronegative, HSV-2 seropositive and who presented to the study clinic with a new genital ulcer. Intention to treat analysis was used.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Acyclovir | Placebo
Number analyzed (Participants) | 61 | 27
Days | 5.1 (0.3) | 6.0 (0.6)

2. Secondary Outcome: Time to First Negative Herpes Simplex Virus (HSV) DNA PCR
Description: To examine the time to first negative HSV DNA PCR among women who have a history of GUD and are HSV-2 seropositive and HIV-1 seronegative, and who are randomized to 400mg acyclovir or matching placebo
Time Frame: Days 1-5, 7, 9, 11, 13
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | Acyclovir | Placebo
Number analyzed (Participants) | 61 | 27
Days | 3.0 (0.3) | 5.0 (0.8)

ADVERSE EVENTS:
Arm/Group | Acyclovir | Placebo
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/27
Other Adverse Events (participants affected / at risk) | 0/61 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No